CLINICAL TRIAL: NCT03228940
Title: An Open-Label Study to Assess the Safety and Effect on Key Biomarkers of Oral RVX000222 in Subjects With Fabry Disease
Brief Title: Safety and Effect of Oral RVX000222 in Subjects With Fabry Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changed development priorities
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVX222-CS-020
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
Keywords: Cardiovascular Disease, Renal Disease
MeSH Terms: conditions — Fabry Disease; Cardiovascular Diseases; Kidney Diseases | interventions — apabetalone

STUDY DESIGN:
Intervention Model Description: Open-label exploratory
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- treatment (Experimental): RVX000222 (apabetalone) 100 mg to be administered orally BID 12 hours apart.
  Interventions: Drug: RVX000222

INTERVENTIONS:
Drug: RVX000222 — oral, BID
  Other Names: apabetalone; RVX-208

SUMMARY:
Fabry Disease (FD) is a rare X-linked lysosomal storage disorder (LSD) caused by mutations in the GLA gene which translates into decreased activity or lack of function of the enzyme alpha-galactosidase A (α-GAL A) and accumulation of the enzymes substrate, i.e., Gb3, throughout the body. Cardiovascular and renal complications are among the leading causes of death in FD patients. RVX000222 is a BET inhibitor which modulates the expression of a variety of genes and, due to its effects on pathways downstream of substrate accumulation and reduction of major cardiac events, holds promise as a potential add-on therapy to accompany enzyme replacement therapy (ERT) in FD patients.

DETAILED DESCRIPTION:
Fabry Disease (FD) is a rare X-linked lysosomal storage disorder (LSD) caused by mutations in the GLA gene coding for the enzyme alpha-galactosidase A (α-GAL A). As a consequence globotriaosylceramide (Gb3), the enzyme's substrate, is not metabolized efficiently. The result is progressive accumulation of Gb3 and related glycosphinglolipids, particularly in blood vessels of the skin, kidney, heart and brain, causing severe complications such as cardiomyopathy, left ventricular hypertrophy and other cardiovascular related issues, as well as renal failure and end stage renal disease, ischemic stroke and peripheral neuropathy.

RVX000222 is a BET inhibitor which modulates the expression of a variety of genes; in a number of Phase 1 and 2 clinical trials RVX000222 significantly affected markers of cardiovascular disease (CVD), such as high-sensitivity C-reactive protein (hs-CRP), alkaline phosphatase, components of the complement and coagulation cascades, and markers of reverse cholesterol transport in patients with CVD. Due to its beneficial effects on several pathways downstream of Gb3 accumulation and MACE reduction, RVX000222 holds promise as a potential add-on therapy to accompany enzyme replacement therapy (ERT) in FD patients. In addition to regulating disease related pathways, RVX000222 treatment significantly affects putative markers associated with FD such as Afamin and intercellular and vascular adhesion molecules in cell cultures.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria may be enrolled:

1. Provide written informed consent before participation in the study.
2. Aged between 18 and 75 years, inclusive.
3. Diagnosis of Fabry disease, either

   1. receiving enzyme replacement therapy for at least 6 months at time of screening (Cohort 1).
   2. not receiving enzyme replacement therapy at time of screening and not having received enzyme replacement therapy in the past (Cohort 2).
4. Female subjects must meet one of the following:

   1. If of childbearing potential, must have a negative urine pregnancy test and must also be willing to practice total abstinence or to use an approved (non-hormonal) form of birth-control throughout the study treatment phase and up to 28 days after the last study drug dose.

      -OR-
   2. Meet at least one of the following criteria:

      * Be postmenopausal, defined as having been amenorrheic for at least 2 years.
      * Have had a hysterectomy or a bilateral oophorectomy.
5. Male subjects who have not had a vasectomy must practice abstinence or use an approved method of birth control, including barrier contraception, throughout the study treatment phase and up to 3 months after the last study drug dose.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled:

1. Patients with stage 5 Chronic Kidney Disease (CKD) receiving renal replacement therapy with either hemodialysis or peritoneal dialysis, renal transplant or with eGFR <15 ml/min/1.73m2.
2. Patients with prior transplantations of organs or bone marrow.
3. Patients with unstable cardiac condition including heart attack, stroke, uncontrolled atrial fibrillation or a major cardiac procedure within 3 months.
4. Current or recent (within 12 months prior to Screening) treatment with cyclosporine.
5. History of malignancy of any organ system, treated or untreated, within the past 2 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
6. Evidence of cirrhosis from liver imaging or biopsy, a history of hepatic encephalopathy, esophageal or gastric varices, active hepatitis, or prior porta-caval shunt procedure, or a Child-Pugh score of at least 5 points.
7. Have a screening 12-lead ECG considered clinically significant by the investigator requiring a corrective intervention in the short-term.
8. Have any known allergy or intolerance to any compound in the test products or any other closely related compound.
9. ALT or AST >1.5 x ULN at Screen.
10. Total bilirubin >ULN at Screen.
11. Use of diclofenac, clavulanic acid or regular use of acetaminophen >1g per day.
12. Have participated in a clinical study and received any investigational medication within the last 30 days preceding Visit 1 (Screening).
13. Patients whose safety may be compromised by study participation due to, for example, an infection within the last 30 days.
14. Are not, in the opinion of the investigator, able or willing to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-22 (Estimated); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | 16 weeks
  Adverse events in Fabry Disease patients from the screening visit until 2 weeks after treatment completion with RVX000222.
Changes in clinical laboratory parameters | 12 weeks
  Changes in chemistry and hematology laboratory test results in Fabry Disease patients throughout and at the end of treatment phase with RVX000222 relative to baseline test results.

SECONDARY OUTCOMES:
Change in Alkaline Phosphatase | 12 weeks
  Change in serum alkaline phosphatase in Fabry Disease patients throughout and at the end of treatment phase with RVX000222 relative to baseline level.
Changes in key markers of Chronic Kidney Disease-Bone Mineral Disease (CKD-BMD) | 12 weeks
  Changes in key markers of CKD-BMD i.e. RANKL and osteoprotegerin in Fabry Disease patients throughout and at the end of treatment phase with RVX000222 relative to baseline levels.
Changes in key markers of inflammation | 12 weeks
  Changes in key markers of inflammation i.e. high-sensitivity C-Reactive Protein (hsCRP) in Fabry Disease patients throughout and at the end of treatment phase with RVX000222 relative to baseline levels.
Changes in markers of alpha-galactosidase (a-GAL A) deficiency | 12 weeks
  Changes in key markers of a-GLA A deficiency i.e. Gb3 and lyso-Gb3 in Fabry Disease patients throughout and at the end of treatment phase with RVX000222 relative to baseline level.
Initial uptake and steady-state level of RVX000222 | 12 weeks
  RVX000222 blood concentration at 4 hours after initial administration in comparison to baseline. Steady-state concentration of RVX000222 and its two principal metabolites, RVX000288 and RVX000404, throughout and at the end of treatment phase with RVX000222.

CONTACTS AND LOCATIONS:
Overall Officials: Michael West, MD, Principal Investigator — Queen Elizabeth II Health Sciences Centre, Victoria General Site
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Victoria General Site, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided